CLINICAL TRIAL: NCT00636155
Title: A Phase II Study of EL625 in Patients in Persistent Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: EL625 in Persistent Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding
Sponsor: David Rizzieri (Other)
Collaborators: Eleos, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David Rizzieri, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001363
Record Dates: First submitted 2008-01-22; First posted 2008-03-14 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Lymphoma, Small Lymphocytic; Leukemia, Lymphocytic, Chronic
Keywords: Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; EL625; cenersen
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients (Experimental): EL625 combined with traditional chemotherapy (rituximab, fludarabine, and cyclophosphamide)
  Interventions: Drug: cenersen sodium; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: cenersen sodium — 2.4 mg/kg/day as a continuous infusion over 24 hours starting on day one and ending on day 4
  Other Names: EL625
Drug: Rituximab — 375 mg/m2 on day 2
  Other Names: Rituxan
Drug: Cyclophosphamide — 250 mg/m2 on days 2, 3, and 4
  Other Names: Cytoxan
Drug: Fludarabine — 25 mg/m2 on days 2, 3, and 4
  Other Names: Fludara

SUMMARY:
The purpose of this research study is to see if the investigational drug EL625, when combined with traditional chemotherapy (rituximab, fludarabine, and cyclophosphamide), is effective in Persistent Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL)

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) and small B-cell lymphocytic lymphoma (SLL) are thought to be different manifestations of the same disease. Treatment options for CLL/SLL range from a watch and wait approach to bone marrow transplant. Currently there is no consensus on the best treatment regimen and new approaches to treatment are needed.

EL625 is a 20-mer antisense molecule which binds to a coding region of exon 10 in p53 RNA transcripts. It can bind to both mutant and wild type p53. p53 is involved in regulating apoptosis and DNA repair in cells. When genetic damage occurs p53 is upregulated. As the expression of p53 increases in normal cells they are more likely to undergo apoptosis rather than cell cycle arrest and DNA repair. However in malignant cells, for a given level of DNA damage they are more likely to undergo cell cycle arrest and repair rather than apoptosis. Because EL625 is theorized to increase response to chemotherapy, we propose adding EL625 to a combination of fludarabine, cyclophosphamide and rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of CLL/SLL who have received at least one prior treatment regimen and have persistent disease (i.e. any evidence of active disease). Patients with a chromosome 17 abnormality or a p53 mutation of any type may be enrolled without having received prior treatment.
* Patients must be 18 years of age or older.
* Patient has an estimated or measured creatinine clearance ≥30 ml/min at study enrollment.
* AST, ALT, total bilirubin < than 2.5 times the upper limit of normal.
* WBC > 1.5; ANC >500; Plt >50,000 unless documented as due to disease
* ECOG performance status of 0-2.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for 2 weeks after administration of the study drug.
* Male subject agrees to use an acceptable method for contraception for the duration of the study therapy and for 2 weeks after administration of study drug.

Exclusion Criteria:

* Female who is pregnant or lactating.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with another malignancy within the last three years (from documentation of remission) other than basal or squamous cell skin cancer, resected early stage prostate cancer not requiring systemic treatment or CIS of the cervix or fully treated early stage prostate cancer.
* Significant cardiac or vascular events within 6 months: acute MI, unstable angina, severe peripheral vascular disease (ischemic pain at rest class 3 or worse, non-healing ulcers/wounds, congestive heart failure (NYHA class ≥ 2), uncontrolled cardiac arrhythmias, and disseminated intravascular coagulation.
* Patients who are unable to refrain from taking acetaminophen
* Investigational agent within 14 days of enrolling on the study.
* Patients unable or unwilling to refrain from antioxidants including vitamin A, vitamin C, vitamin E, lycopene, lutein, grape seed extract, pycnogenol, green tea extract, and the like.
* Patients who have received a prior allogenic stem cell transplant and have at least 2.5% donor cells still evident on engraftment studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled from Duke University Medical Center.
Groups:
- All Patients: EL625 2.4mg/kg/day as a continuous infusion daily for 4 days combined rituximab 375mg/m2 IV on day 2, fludarabine IV 25mg/m2 over 30 minutes on days 2- 4 and cyclophosphamide IV 250mg/m2 over 1 hour on days 2-4.
Period: Overall Study
Arm/Group | All Patients
Started | 20
Completed | 2 (Completed maximum 6 cycles of treatment)
Not Completed | 18
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 3
Not completed — Stem cell transplant | 1
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age Continuous [Median (Full Range); unit: years] | 62 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Overall Response (Complete Response + Partial Response)
Description: Overall Response is the total number of participants with a Complete (CR) or Partial (PR) response. CR requires the absence of lymphadenopathy, hepatomegaly or splenomegaly and constitutional symptoms and a normal CBC; bone marrow must be at least normocellular for age, with less than 30% nucleated cells being lymphocytes with no lymphoid nodules. Partial Response: requires ≥ 50% decrease in one of the following: peripheral blood lymphocyte count, lymphadenopathy, enlargement of liver and/or spleen, or bone marrow involvement by CLL AND at least one hematologic parameter met for 2 months.
Time Frame: every 3 cycles
Population: Patients completing at least 2 cycles of treatment
Measure: Number; unit: participants
Groups:
- All Patients: Patients treated with cenersen, fludarabine, cyclphosphamide and rituximab
Arm/Group | All Patients
Number analyzed (Participants) | 17
participants | 9

2. Secondary Outcome: Progression Free Survival
Description: Progression is defined as at least one of the following: 1) ≥ 50% increase in the sum of the products of at least two lymph nodes one two consecutive determinations (at least one node must be ≥ 2 cm); appearance of new palpable lymph nodes, 2) ≥ 50% increase in the size of the liver and/or spleen; appearance of palpable hepatomegaly or splenomegaly, which was not previously present, 3) ≥ 50% increase in the absolute number of circulating lymphocytes to at least 5,000/µl or 4)Transformation to a more aggressive histology.
Time Frame: 5 years
Population: All patients who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 20
months | 5.3 [4.7 to 14.0]

3. Secondary Outcome: Overall Survival
Time Frame: 5 years
Population: All patients who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 20
months | 10.6 [5.37 to NA] — The upper limit of the confidence interval has not been reached/insufficient number of participants

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of study treatment until 30 days after the last dose.
Description: Other AE section contains all AEs, including SAEs, regardless of attribution to study drug
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=20)
Neutrophils / granulocytes (ANC / AGC) (Investigations) | 1 (1)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 3 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=20)
Allergic reaction / hypersensitivity (including drug fever) (Immune system disorders) | 2 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergy / Immunology - Other (Immune system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 10 (16)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (2)
Leukocytes (total WBC) (Investigations) | 8 (13)
Neutrophils / granulocytes (ANC / AGC) (Investigations) | 6 (7)
Platelets (Investigations) | 14 (16)
Palpitations (Cardiac disorders) | 2 (2)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (3)
Supraventricular and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 2 (2)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 (1)
Cardiac General - Other (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (5)
INR (International Normalized Ratio of prothrombin time (Investigations) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 11 (15)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9/L) (General disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (7)
Rigors / chills (General disorders) | 5 (6)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 4 (4)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 3 (3)
Dermatology / Skin - Other (Skin and subcutaneous tissue disorders) | 5 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hair Loss / Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus / itching (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Atrial flutter (Cardiac disorders) | 1 (1)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 5 (5)
Ulceration (Skin and subcutaneous tissue disorders) | 3 (3)
Hot flashes / flushes (Vascular disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dysphagia (difficulty swallowing (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis / stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (10)
Obstruction, GI - Ileum (Gastrointestinal disorders) | 1 (1)
Taste Alteration (dysgeusia) (Nervous system disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hemorrhage / Bleeding - Other (Vascular disorders) | 1 (1)
Hemorrhage, GU - Kidney (Renal and urinary disorders) | 2 (2)
Petechiae / purpura (hemorrhage / bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1)
Liver dysfunction / failure (clinical) (Hepatobiliary disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin w/oclinically or microbiologically documented infe (Blood and lymphatic system disorders) | 7 (9)
Infection - Other (Infections and infestations) | 3 (4)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Bladder (urin (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils-Lip / perioral (Infections and infestations) | 1 (2)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Rectum (Infections and infestations) | 2 (2)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Urinary tract (Infections and infestations) | 1 (1)
Dermal change lymphedema, phlebolymphedema (Vascular disorders) | 3 (3)
Edema: limb (General disorders) | 4 (5)
Edema: pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (4)
Alkaline phosphatase (Investigations) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 2 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (6)
Creatinine (Investigations) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (10)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (3)
Metabolic / Laboratory - Other (Investigations) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (4)
Uric Acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (2)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body / generalized (Musculoskeletal and connective tissue disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (7)
Memory Impairment (Nervous system disorders) | 2 (2)
Mood Alteration - Agitation (Psychiatric disorders) | 1 (2)
Mood Alteration - Anxiety (Psychiatric disorders) | 3 (3)
Mood Alteration - Depression (Psychiatric disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Psychosis (hallucinations / delusions) (Psychiatric disorders) | 2 (2)
Somnolence / depressed level of consciousness (Nervous system disorders) | 1 (2)
Syncope (fainting) (Nervous system disorders) | 2 (2)
Dry Eye Syndrome (Eye disorders) | 1 (1)
Vision - blurred vision (Eye disorders) | 3 (3)
Musculoskeletal - Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Dental / teeth / peridontal (Gastrointestinal disorders) | 1 (1)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Head / headache (Nervous system disorders) | 6 (6)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Lymph node (Blood and lymphatic system disorders) | 1 (1)
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain - Other (General disorders) | 1 (1)
Pulmonary / Upper Respiratory - Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary / Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Urinary frequency / urgency (Renal and urinary disorders) | 5 (6)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No